CLINICAL TRIAL: NCT02509936
Title: Crowd Funding and Social Networks as a Novel Mechanism to Promote Sustainable Physical Growth and Positive Psychosocial and Neurodevelopmental Outcomes in Severely Stunted Guatemalan Children
Brief Title: Promoting Physical Growth and Positive Development in Severely Stunted Guatemalan Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuqu' Kawoq, Maya Health Alliance (Other)
Collaborators: Universidad del Valle, Guatemala (Other); Grand Challenges Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WK-2015-003
Record Dates: First submitted 2015-07-17; First posted 2015-07-28 (Estimated); Results first posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Malnutrition; Developmental Disabilities
MeSH Terms: conditions — Malnutrition; Developmental Disabilities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care Arm (Active Comparator): In this arm enrolled children will receive the national standard of care for growth support, which includes growth monitoring, a food ration, and a multiple micronutrient powder supplement.
  Interventions: Dietary Supplement: Standard-of-care nutrition support
- Home-based Education (Experimental): In the intervention arm, children will receive the national standard of care for growth support, which includes growth monitoring, a food ration, and a multiple micronutrient powder supplement. In addition, they will receive monthly home visits from a community health promoter who will provide detailed dietary assessments and individualized dietary coaching and education to parents.
  Interventions: Behavioral: Home-based nutrition education; Dietary Supplement: Standard-of-care nutrition support

INTERVENTIONS:
Behavioral: Home-based nutrition education — Health promoters will use 24-hour dietary recall information to assess meal frequency and dietary diversity and then provide tailored nutrition coaching to parents.
  Arms: Home-based Education
Dietary Supplement: Standard-of-care nutrition support — Subjects will be provided with a standard food ration and with a multiple micronutrient powder dietary supplement (Chispitas)

SUMMARY:
This study seeks to evaluate the impact of an intensive home-based education intervention targeting severely stunted Guatemalan children for catch up growth and improved development. Half of the children in the study will receive standard of care, which includes micronutrient supplementation and a food ration. The other half of children in the study will receive, in addition to the above, home-based dietary assessment and individualized parental nutrition education.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 6-24 months at time of enrollment
* Height/length for age Z score of less than -2.5
* Child lives with parent/legal guardian

Exclusion Criteria:

* Presence of acute malnutrition (weight for length/height Z score of less than -2)
* Presence of other severe medical illness (e.g. congenital heart disease, genetic abnormality)

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 324 (Actual)
Dates: Start 2015-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rohloff, MD PhD, Principal Investigator — Wuqu' Kawoq; Maria Grazioso, PhD, Principal Investigator — Universidad del Valle, Guatemala
Locations (1):
- Wuqu' Kawoq, Tecpán Guatemala, Departamento de Chimaltenango, Guatemala

REFERENCES:
- [Derived] Martinez B, Cardona S, Rodas P, Lubina M, Gonzalez A, Farley Webb M, Grazioso MDP, Rohloff P. Developmental outcomes of an individualised complementary feeding intervention for stunted children: a substudy from a larger randomised controlled trial in Guatemala. BMJ Paediatr Open. 2018 Oct 3;2(1):e000314. doi: 10.1136/bmjpo-2018-000314. eCollection 2018. PMID 30306144
- [Derived] Martinez B, Webb MF, Gonzalez A, Douglas K, Grazioso MDP, Rohloff P. Complementary feeding intervention on stunted Guatemalan children: a randomised controlled trial. BMJ Paediatr Open. 2018 Apr 27;2(1):e000213. doi: 10.1136/bmjpo-2017-000213. eCollection 2018. PMID 29719876

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care Arm: In this arm enrolled children received the national standard of care for growth support, which includes growth monitoring, a food ration, and a multiple micronutrient powder supplement.
  Standard-of-care nutrition support: Subjects were provided with a standard food ration and with a multiple micronutrient powder dietary supplement (Chispitas)
- Home-based Education: In the intervention arm, children received the national standard of care for growth support, which includes growth monitoring, a food ration, and a multiple micronutrient powder supplement. In addition, they received monthly home visits from a community health promoter who provided detailed dietary assessments and individualized dietary coaching and education to parents.
  Home-based nutrition education: Health promoters used 24-hour dietary recall information to assess meal frequency and dietary diversity and then provide tailored nutrition coaching to parents.
  Standard-of-care nutrition support: Subjects were provided with a standard food ration and with a multiple micronutrient powder dietary supplement (Chispitas)
Period: Overall Study
Arm/Group | Standard of Care Arm | Home-based Education
Started | 163 | 161
Completed | 151 | 145
Not Completed | 12 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care Arm | Home-based Education | Total
Number analyzed (Participants) | 163 | 161 | 324
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 163 | 161 | 324
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 15.1 (5.2) | 15.8 (5.2) | 15.4 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 69 | 142
  Male | 90 | 92 | 182
Region of Enrollment [Number; unit: participants]
  Guatemala | 163 | 161 | 324
Weight for age Z score [Mean (Standard Deviation); unit: Z score] — A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Higher values above zero are indicative of higher than normal weight for age. Lower values below zero are indicative of lower than normal weight for age.
  Z score | -1.92 (0.79) | -1.95 (0.76) | -1.93 (0.77)
Length/height for age [Mean (Standard Deviation); unit: Z score] — A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Higher values above zero are indicative of higher than normal length/height for age. Lower values below zero are indicative of lower than normal length/height for age.
  Z score | -3.41 (0.74) | -3.47 (0.73) | -3.43 (0.73)

OUTCOME MEASURES:

1. Primary Outcome: Change in Height/Length for Age Z Score
Description: Change in height/length over 6 months. Tool used is the WHO Child Growth Reference Standards. Change values calculated as: 6 month (z-score) minus Baseline (z-score).
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: Z scores
Arm/Group | Standard of Care Arm | Home-based Education
Number analyzed (Participants) | 151 | 145
Z scores | -0.02 (0.45) | 0.05 (0.48)

2. Secondary Outcome: Cognitive Development
Description: Change in cognitive development Z score over 6 months. Tool used: Bayley III Cognitive Development Observational Checklist. Z-scores derived internally from the entire baseline measurement data set for the study. A z-score of 0 is equal to the mean cognitive score for the study population at baseline. Lower numbers indicate values lower than the baseline study population mean mean and higher numbers indicate values higher than this mean. Higher values above zero are indicative of cognitive scores higher than mean baseline score for the study population. Lower values below zero are indicative of cognitive scores lower than mean baseline score for the study population. For outcomes, change values are calculated as 6 month (z-score) minus Baseline (z-score)
Time Frame: Baseline, 6 months
Population: Due to expense constraints, a subset of subjects (consecutively recruited during the first 5 months (n=210 enrolled vs. 324 enrolled in study overall)) were invited to participate in the psychometric substudy. Subsequently, only 147 completed both time point assessments, and 47 were excluded for aging-out of the Z score internal reference norms.
Measure: Mean (95% Confidence Interval); unit: Z score
Arm/Group | Standard of Care Arm | Home-based Education
Number analyzed (Participants) | 53 | 47
Z score | 0.38 [0.05 to 0.72] | 0.28 [-0.14 to 0.71]

3. Secondary Outcome: Socioemotional Development
Description: Change in socioemotional development score over 6 months. Tool used: Bayley III Socioemotional Development Parent Questionnaire. Z-scores derived internally from the entire baseline measurement data set for the study. A z-score of 0 is equal to the mean socioemotional score for the study population at baseline. Lower numbers indicate values lower than the baseline study population mean mean and higher numbers indicate values higher than this mean. Higher values above zero are indicative of socioemotional scores higher than mean baseline score for the study population. Lower values below zero are indicative of socioemotional scores lower than mean baseline score for the study population. For outcomes, change values are calculated as 6 month (z-score) minus Baseline (z-score)
Time Frame: Baseline, 6 months
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Z score
Arm/Group | Standard of Care Arm | Home-based Education
Number analyzed (Participants) | 53 | 47
Z score | 0.44 [0.07 to 0.81] | 0.20 [-0.13 to 0.53]

4. Secondary Outcome: Gross Motor Development
Description: Change in gross motor development score over 6 months. Tool used: Bayley III Gross Motor Observational Checklist. Z-scores derived internally from the entire baseline measurement data set for the study. A z-score of 0 is equal to the mean gross motor score for the study population at baseline. Lower numbers indicate values lower than the baseline study population mean mean and higher numbers indicate values higher than this mean. Higher values above zero are indicative of gross motor scores higher than mean baseline score for the study population. Lower values below zero are indicative of gross motor scores lower than mean baseline score for the study population. For outcomes, change values are calculated as 6 month (z-score) minus Baseline (z-score)
Time Frame: Baseline, 6 months
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Z score
Arm/Group | Standard of Care Arm | Home-based Education
Number analyzed (Participants) | 53 | 47
Z score | 0.51 [0.18 to 0.85] | 0.70 [0.3 to 1.1]

5. Secondary Outcome: Fine Motor Development
Description: Change in fine motor development score over 6 months. Tool used: Bayley III Fine Motor Observational Checklist. Z-scores derived internally from the entire baseline measurement data set for the study. A z-score of 0 is equal to the mean fine motor score for the study population at baseline. Lower numbers indicate values lower than the baseline study population mean mean and higher numbers indicate values higher than this mean. Higher values above zero are indicative of fine motor scores higher than mean baseline score for the study population. Lower values below zero are indicative of fine motor scores lower than mean baseline score for the study population. For outcomes, change values are calculated as 6 month (z-score) minus Baseline (z-score)
Time Frame: Baseline, 6 months
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Z score
Arm/Group | Standard of Care Arm | Home-based Education
Number analyzed (Participants) | 53 | 47
Z score | 0.27 [-0.09 to 0.63] | 0.4 [0.04 to 0.76]

6. Secondary Outcome: Receptive Language Development
Description: Change in receptive language development score over 6 months. Tool used: Bayley III Receptive Language Observational Checklist. Z-scores derived internally from the entire baseline measurement data set for the study. A z-score of 0 is equal to the mean receptive language score for the study population at baseline. Lower numbers indicate values lower than the baseline study population mean mean and higher numbers indicate values higher than this mean. Higher values above zero are indicative of receptive language scores higher than mean baseline score for the study population. Lower values below zero are indicative of receptive language scores lower than mean baseline score for the study population. For outcomes, change values are calculated as 6 month (z-score) minus Baseline (z-score)
Time Frame: Baseline, 6 months
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Z score
Arm/Group | Standard of Care Arm | Home-based Education
Number analyzed (Participants) | 53 | 47
Z score | 0.56 [0.21 to 0.92] | 0.49 [0.11 to 0.86]

7. Secondary Outcome: Expressive Language Development
Description: Change in expressive language development score over 6 months. Tool used: Bayley III Expressive Language Observational Checklist. Z-scores derived internally from the entire baseline measurement data set for the study. A z-score of 0 is equal to the mean expressive language score for the study population at baseline. Lower numbers indicate values lower than the baseline study population mean mean and higher numbers indicate values higher than this mean. Higher values above zero are indicative of expressive language scores higher than mean baseline score for the study population. Lower values below zero are indicative of expressive language scores lower than mean baseline score for the study population. For outcomes, change values are calculated as 6 month (z-score) minus Baseline (z-score)
Time Frame: Baseline, 6 months
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Z score
Arm/Group | Standard of Care Arm | Home-based Education
Number analyzed (Participants) | 53 | 47
Z score | 0.63 [0.34 to 0.93] | 0.69 [0.38 to 0.99]

8. Secondary Outcome: Minimum Diet Diversity
Description: Number of participants meeting the age appropriate minimum number of food groups consumed per day. This is defined according to the WHO's Infant and Young Child Feeding Indicators guidelines as greater or equal to 4 food groups consumed in the last 24 - hour period. The 7 possible food groups are: (1) grains, roots, tubers; (2) legumes, nuts; (3) dairy products; (4) flesh foods; (5) eggs; (6) vitamin A-rich fruits and vegetables; (7) other fruits and vegetables.
Time Frame: 0 months, 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Arm | Home-based Education
Number analyzed (Participants) | 151 | 145
Participants | 115 | 135

9. Secondary Outcome: Minimum Meal Frequency
Description: Number of participants meetings the age-appropriate number of solid meals per day. This is defined according to the WHO's Infant and Young Child Feeding Indicators guidelines as 2 solid meals in the last 24-hour period for breastfed infants 6-8 months old; 3 solid meals in the last 24-hour period for breastfed infants 9 months or older; 4 solid meals in the last 24-hour period for non-breastfed infants.
Time Frame: 0 months, 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Arm | Home-based Education
Number analyzed (Participants) | 151 | 145
Participants | 131 | 129

10. Secondary Outcome: Minimum Acceptable Diet
Description: Number of participants who meet both minimum diet diversity and minimum meal frequency indicators. Minimum diet diversity and minimum meal frequency are both defined according to the WHO's Infant and Young Child Feeding Indicators guidelines. See the entries for minimum diet diversity and minimum meal frequency in this record for more details.
Time Frame: 0 months, 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Arm | Home-based Education
Number analyzed (Participants) | 151 | 145
Participants | 104 | 123

ADVERSE EVENTS:
Arm/Group | Standard of Care Arm | Home-based Education
Serious Adverse Events (participants affected / at risk) | 0/163 | 0/161
Other Adverse Events (participants affected / at risk) | 0/163 | 0/161

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No